CLINICAL TRIAL: NCT04684121
Title: A Phase 2, Prospective, Randomized, Double-Blind, Parallel-Group, Within-Subject Vehicle Controlled Multicenter Study of the Efficacy and Safety of Granexin® Gel to Improve Burn Wound Healing
Brief Title: Study of the Efficacy and Safety of Granexin® Gel to Improve Burn Wound Healing
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No longer aligned with company strategy
Sponsor: Xequel Bio, Inc. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-BURN-01; CDMRP-MB190074 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2020-12-17; First posted 2020-12-24 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Second Degree Burn; Thermal Burn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Granexin gel (Experimental): Within-subject comparison of Granexin® Gel versus vehicle gel (placebo).
  Granexin® gel 200 μM will be applied daily over ten days. Granexin® will be applied to one of two selected target burns.
  Interventions: Drug: Granexin® gel (200 μM)
- Vehicle Gel (Placebo Comparator): Within-subject comparison of Granexin® Gel versus vehicle gel (placebo).
  Vehicle gel will be applied daily over ten days. Vehicle will be applied to one of two selected target burns.
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: Granexin® gel (200 μM) — Granexin® gel (200 μM) will be topically applied once daily for 10 days in association with standard of care (SOC) wound cleaning and ACTICOAT Flex 3TM dressing.
  Arms: Granexin gel
Drug: Vehicle gel — Vehicle gel will be topically applied once daily for 10 days in association with standard of care (SOC) wound cleaning and ACTICOAT Flex 3TM dressing.
  Arms: Vehicle Gel

SUMMARY:
To evaluate the efficacy of Granexin® gel to promote accelerated healing of second-degree (deep partial thickness) thermal burns.

DETAILED DESCRIPTION:
Multi-center, prospective, randomized, double-blind, parallel-group, within-subject Vehicle controlled, safety and efficacy trial involving subjects with two comparable (similar body location, similar burn area and burn severity), noncontiguous deep second-degree thermal burns of less than 20% TBSA. A total of 30 subjects will have two target burns randomly assigned in a ratio of 1:1 to two treatment groups.

* Granexin® gel (200 μM) plus ACTICOAT Flex 3TM
* Vehicle gel plus ACTICOAT Flex 3TM

The study procedures are divided into the following three periods:

* Screening (within 36 hours of the time of injury)
* Treatment (daily for 10 days)
* Follow-up (Day 10 through Month 12)

The anticipated total duration of a given subject's participation in this study is 12 months. Screening can occur up to 36 hours prior to Day 0; Screening and Day 0 may occur on the same day. Treatment period visits occur daily from Day 0 through Day 9, on-site and remotely. During the treatment period, each subject will be treated with Granexin® gel (200 μM) plus ACTICOAT Flex 3TM on one target burn and Vehicle gel plus ACTICOAT Flex 3TM on the second target burn. After Day 9, the subject will return to clinic on Day 10 and be followed-up (on-site or remotely) every other day thereafter until Day 28, with on-site visits on Days 14, 20, and 28. The subject will then return to the clinic for follow-up visits at Months 6, 9, and 12.

Safety will be assessed during the study by monitoring adverse events and measuring vital signs at each on-site visit, electrocardiograms (ECG), and clinical laboratory tests at selected time points before and after treatment with Granexin® gel and Vehicle gel. Concomitant medications will be reviewed at every visit.

ELIGIBILITY:
Subjects will be eligible for randomization in the study if they meet all of the following inclusion criteria:

1. Aged 18 years or older
2. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and must agree to use hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence from the time of informed consent through Day 28 of the study; or female subjects must be postmenopausal (defined as 12 months since last menstruation) or surgically sterilized.

   Male subjects must abstain from sex with WOCBP or use an adequate method of contraception (as described above) from the time of informed consent through Day 28 of the study.
3. Must have two comparable (similar body location, similar burn area and burn severity), noncontiguous deep second-degree thermal burns (target burns) caused by a fire/flame, scalds, or a hot object.
4. Must have two target burns:

   1. No single target burn less than 1% TBSA
   2. All burns less than 20% cumulative TBSA
5. Any treatment administered prior to randomization must be similar to both target burns and must be removed or discontinued prior to randomization.
6. Signed informed consent form

Subjects will not be eligible for randomization in the study if any of the following exclusion criteria are met:

1. Chemical, radiation, or electrical burns
2. Burns older than 36 hours prior to study randomization
3. Target burns more severe than deep second-degree
4. Target burns to the hands, face, neck, or feet. Burn area may include hands and feet where target burn will only include areas extending above the wrist or ankle.
5. Target burns that are superficial second-degree burn wounds expected to heal within two weeks
6. Evidence of active infection, including cellulitis, at the site of the target burns
7. Known collagen vascular diseases
8. Any history of malignancy within the last 5 years or the presence of any active systemic cancer (exception will be basal cell skin cancer in a non-burned area)
9. History of clinically significant cardio/pulmonary conditions
10. Clinically significant medical conditions as determined by the clinical Investigator, which would impair wound healing including renal, hepatic, hematologic, neurologic, or immune disease
11. Known inability or unavailability to complete required study visits
12. Critical illnesses such as those requiring ventilator support, or having a systemic infection or hemodynamic instability, defined as a mean arterial pressure less than 60 mm Hg or requiring vasoactive medications to support blood pressure
13. Major acute or chronic medical illnesses that could affect wound healing (e.g. peripheral vascular disease, insulin dependent diabetes, blood clotting disorder)
14. Currently receiving treatment with medications that inhibit or compromise wound healing. Examples include immunosuppressive agents, topical growth factors, therapeutic anticoagulants, antiplatelet drugs, and systemic steroids such as warfarin, clopidogrel, or prednisone. The use of anticoagulants does not include deep vein thrombosis (DVT) prophylaxis. Subjects may use aspirin or lovenox.
15. Any condition which, in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study
16. Clinically relevant serious co-morbid medical conditions including, but not limited to: unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled cardiac arrhythmias, chronic obstructive or chronic restrictive pulmonary disease, active central nervous system (CNS) disease uncontrolled by standard of care
17. Known positive status for human immunodeficiency virus (HIV), or active hepatitis B or C, or cirrhosis
18. Psychiatric illness/social situations that would limit compliance with study requirements
19. Pregnant or breastfeeding
20. Treatment with another investigational drug within 30 days or 5 half-lives of drug prior to Screening, whichever is longer
21. Known hypersensitivity to the ingredients in Granexin® or ACTICOAT Flex 3TM
22. Known hypersensitivity or allergy to silver or polyester
23. Any other factor, which may, in the opinion of the Investigator, compromise participation and follow-up in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Time to re-epithelization | From Day 0 to Month 12
  Time (in days) to 100% re-epitheliazation of deep second degree burns as determined through clinical assessments

SECONDARY OUTCOMES:
Reduction in scar severity at Month 12 | Month 12
  Assessed using the Vancouver Scar Scale. The Vancouver Scar Scale has 4 variables: Vascularity, Height (thickness), Pliability, Pigmentation. Each variable has three to six possible scores. The scores for the four components will be added to obtain the total score. The total score ranges from 0 to 13, whereby a score of 0 reflects normal skin.
Proportion of burns that convert from partial thickness burns to full thickness burns | From Day 0 to Day 28
  Burn conversion is determined through clinical assessment.
Proportion of subjects needing additional burn interventions | From Day 0 to Day 28
  Determined by the initiation of burn interventions, including surgery and skin grafts
Time to skin grafting | From Day 0 to Month 12
  Determined by time (in days) to skin grafting
Incidence of infection | From Day 0 to Month 12
  Determined by Investigator's assessment of presence or absence of infection
Incidence of treatment related adverse events (AEs) | From Day 0 to Month 12
  Assessed using Common Terminology Criteria for Adverse Events (CTCAE) v 5.0. Events that are probably, possible, and definitely related will be considered treatment related events.

OTHER OUTCOMES:
Reduction in scar severity | Months 6 and 9
  Assessed using the Vancouver Scar Scale. The Vancouver Scar Scale has 4 variables: Vascularity, Height (thickness), Pliability, Pigmentation. Each variable has three to six possible scores. The scores for the four components will be added to obtain the total score. The total score ranges from 0 to 13, whereby a score of 0 reflects normal skin.
Histological examination of burns | Punch biopsies collected from each target burn on Day 0, Day 7 and Month 12
  Analysis of punch biopsies taken from the center of each target burn: depth of injury to dermis measured as vertical height (microns) to the most deeply injured area measured from each histologic section, assessment of inflammatory cell infiltration via direct counting of inflammatory cells from each histologic section, scoring of collagen organization from each histologic section.
Exploratory gene expression for markers of wound healing and scar formation | Collected from each target burn on Day 0, Day 7 and Month 12
  Gene expression levels of pharmacodynamic markers of wound healing and scar formation will be evaluated by multiplex direct gene counting assay.

IPD SHARING:
Plan to Share IPD: No